CLINICAL TRIAL: NCT04059354
Title: Down Syndrome Speech Intelligibility Diagnostic Treatment Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Office of the Vice Chancellor for Research and Graduate Education (Unknown); Wisconsin Alumni Research Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019-0706; A348700 (Other: UW Madison); VCRGE/WAISMAN/WAISMAN (Other: UW Madison); Protocol Version 12/10/2019 (Other: UW Madison)
Record Dates: First submitted 2019-08-14; First posted 2019-08-16 (Actual); Results first posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Down Syndrome
Keywords: Speech intelligibility
MeSH Terms: conditions — Down Syndrome; Speech Intelligibility

STUDY DESIGN:
Intervention Model Description: Multiple single-subject design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Speech therapy (Experimental): Treatment: Direct speech therapy will be provided for a 12 week period with up to three one-hour sessions per week (36 sessions per participant) as tolerated and 30 minutes weekly home practice.
  Interventions: Behavioral: Speech therapy addressing phonology and motor learning

INTERVENTIONS:
Behavioral: Speech therapy addressing phonology and motor learning — Determine the efficacy of a newly devised intensive speech treatment plan, to use with individuals with Down syndrome, that combines two treatment approaches: Cycles Phonological Remediation Approach and Script training, while adapting each to prioritize use of practice words with low vowels given research findings that the low vowels /ɑ/ as in 'hot' and /æ/as in 'hat' are less intelligible than the high vowels /i/ as in 'heat' and /u/ as in 'boot'; also, vowel acoustic analyses that revealed word-intelligibility to improve when the production of the low vowels /ɑ/ and /æ/ had more distinctive second formants/vocal tract resonances (a measure that is associated with tongue front-back movement). Each intervention session will include 40-50 minutes of the adapted 'Cycles Phonological Remediation Approach' focusing on articulatory/phonological training at the syllable/word level, and 10-20 minutes of the adapted Script program for motor training at the sentence level.
  Other Names: Speech motor learning

SUMMARY:
The 'Down syndrome speech intelligibility diagnostic treatment study' is a pilot clinical intervention study assessing the efficacy of an integrative speech treatment approach for individuals with Down syndrome (DS). This study will use a single-subject design with 10 male participants with DS, aged 7 to 16 years. The proposed intervention, combines two treatment approaches that are documented to be efficacious with other speech disorders: 1) The Cycles Phonological Remediation Approach, designed for highly unintelligible speech, as guided by the Hodson Assessment of Phonological Patterns (HAPP-3); and 2) Script training, a functional speech motor intervention that promotes phrase-level productions. During the twelve-week intensive intervention period, both approaches will be adapted to prioritize the production of words with low vowels to incorporate increased practice of the low-front and low-back vowels. This modification is based on the investigator's perceptual, acoustic and anatomic research findings. Outcome measures will include perceptual, intelligibility, and acoustic analyses obtained from acoustic recordings. These measures will be used to assess treatment efficacy, and to gain insight into the motoric versus anatomic limitations in speech production commonly present in individuals with DS.

DETAILED DESCRIPTION:
The 'Down syndrome speech intelligibility diagnostic treatment study' is a pilot clinical intervention study assessing the efficacy of an integrative speech treatment approach for individuals with Down syndrome (DS). The clinical management of communication disorders in individuals with DS is a priority for NIH's National Institute on Deafness and Other Communicative Disorder. This priority is well-justified, as DS is a common genetic disorder that causes lifelong intellectual disability where speech intelligibility is typically compromised affecting quality of life.

A number of factors affect speech intelligibility, including difficulties in the production of consonants and vowels. The investigator's research (see references) has identified specific challenges in the production and perception of select vowels, specifically the vowels/æ/ and /ɑ/ (as in hat and hot) that are produced with the tongue in the low/vertical position, with /æ/ in a front horizontal position and /ɑ/ in a back horizontal position. Such findings are indicative of difficulties and/or limitations in regulating tongue height and advancement/retraction likely due to motoric factors and/or craniofacial differences. The DS phenotype commonly includes an underdeveloped midface with maxillary hypoplasia, small hard palate, and relative macroglossia which can restrict tongue movements. Furthermore, the investigator's findings revealed that males are less intelligible than females. Based on Vocal Tract Development Laboratory's (VTLab) research findings on anatomic, acoustic and perceptual studies from speakers with DS (see references), the proposed intervention combines and adapts two well-established speech treatment approaches on articulatory accuracy and motor learning while adapting each approach to prioritize the production of the low-front /æ/ and low-back /ɑ/ vowels over other vowels to provide increased practice in regulating tongue position. The articulatory accuracy treatment uses the Cycles phonological approach designed for highly unintelligible speech, as guided by the Hodson Assessment of Phonological Patterns (HAPP-3); and the motor learning treatment uses Script training using functional common conversational topics with short phrase level productions. Given the wide range of individual differences in individuals with DS, a single-subject design is employed with 10 male participants with DS, aged 7 to 16 years. Each participant will receive a 12-week period of individualized intensive speech-intervention (2-3 hours per week). Data collection will include intake information such as hearing screening, mean length of utterance, receptive vocabulary and oral motor exam. Baseline and outcome measure assessments will follow, comprising perceptual, intelligibility and acoustic analyses derived from acoustic recordings of speech productions (recording and analysis methods similar to procedures described in listed references). Acoustic recordings of the Hodson Assessment of Phonological Patterns-Third Edition (HAPP-3) stimuli will be used for outcome measures 1, 2 and 5; VTLab Speech Production stimuli for outcome measures 3 and 4; and script phrases for outcome measure 6. Finally, the Intelligibility in Context Scale, as rated by parents, for outcome measure 7. An overview of methods for outcome measures data collection follows:

I. The Hodson Assessment of Phonological Patterns-Third Edition (HAPP-3) is a valid, reliable, standardized test designed for children with highly unintelligible speech. It aims to: 1) determine phonological disorder severity (first outcome measure); 2) identify phonological patterns for treatment using the Cycles Phonological Approach (described below, second outcome measure); and 3) track progress through pre- and post- intervention scores (1- and 6-month follow-ups are incorporated in this study design).

The test uses 50 words (32 monosyllabic + 18 multisyllabic) for a comprehensive phonological evaluation to determine the severity of the phonological disorder that impacts communication. In addition, the test categorizes the phonological deviations/errors into two main patterns (omissions and substitutions): 'Word/Syllable Structure Omissions', and 'Consonant Category Deficiencies'. The test offers 129 instances of omissions of: syllables, consonant clusters, or single consonants; and 144 instances of deficiencies/substitutions that include: consonant substitutions and/or assimilations or consonant harmony. Instances of phonological deviations/errors are added, and higher incidence of error pattern/types are targeted first during intervention. The combined total sum of the two phonological deviation patterns (Word/Syllable Omissions Sum plus Consonant Category Deficiencies Sum) yields the Total Occurrences of Major Phonological Deviations (TOMPD) score that is used to determine the severity rating of the phonological disorder in children. Although the total number of Omissions and Deficiencies add up to 273, the TOMPD uses a score range 0-to-150 to rate the severity of the phonological deviation using the following ratings: 0: No errors; 1-50: Mild; 51-100: Moderate; 101-150: Severe; >150: Profound. A decrease in TOMPD score after intervention suggests improvement in speech production/fewer phonological deviations and improved communication/speech intelligibility. A decrease in the sum of the 'Word/Syllable Structure Omissions' and/or the 'Consonant Category Deficiencies' implies fewer errors in that specific pattern of phonological deviation. Furthermore, if the specific type of deviation (omission/substitution) is an intervention target, then the decreased score implicates responsiveness to the Cycles intervention provided (described next). Basically, smaller score/sum indicate fewer errors and higher score/sums reflects more errors/phonological deviations.

The Cycles Phonological Approach is a treatment guidance with focus on assessing and treating speech sound disorders in targeted patterns based on developmental phonology. 'Cycles' refers to periods where all phonological error patterns are facilitated in succession per target phoneme with gradual increase in complexity per cycle. The approach uses a developmental hierarchy of phonological treatment is syllable units, consonant vowel (CV), VC, CVC or VCV, /s/ clusters and alveolars in words, then phrases. The Cycles approach accounts for a number of deficits (such as motoric, phonologic and hearing loss) that are commonly present in individuals with DS. Cycles approach uses production drills and sound practice (i.e. repeating sounds, syllables, & words as practice), in facilitated context to yield accurate productions, where repeat practice may assist with motor control planning (e.g., apraxia, dysarthria). Cycles also uses headphones with amplification, for auditory bombardment of the target sounds, which may assist with hearing loss given likely fluctuating history of otitis media in DS. Adapting the Cycles approach for the proposed treatment plan by prioritizing the low vowels to establish distinct contrasts between /ɑ/ and /æ/, while following the targeted cycles of phonological intervention, adheres to the Cycles program design.

II. The Vocal Tract Development Lab (VTLab) Stimuli were originally designed for lifespan studies of vowel acoustics and included the following considerations: 1) Familiarity to young children; 2) preference to words containing sounds that typically emerge earlier in development, such as bilabial and alveolar consonants versus velars (e.g., 'bat' was chosen over 'cat'); 3) Selection of words with high phonological neighborhood density to maximize vowel acoustic space, an acoustic measure related to speech intelligibility. VTLab stimuli consist of 25 monosyllabic monosyllabic words. Word stimuli include five words for each of the four extreme vowels (/i, u, æ, ɑ/) and the central vowel (/ə/) as in 'eat', 'hoot', 'hat', 'hot', and 'hug' with two of the five words, denoted with the subscript 2, produced twice. The stimuli for the five vowels included the following words: /i/: bead2, eat2, bee, sheep, feet; /u/: boot2, hoot2, boo, shoe, zoo; /æ/: bat2, hat2, bath, cat, sad; /ɑ/: pot2, hot2, top, hop, dot; and /ə/: bug2, hug2, bus, duck, tub. Acoustic recordings of all word stimuli will be used for perceptual and intelligibility assessments. Additionally, the vowel portions of recorded words containing the low vowels /æ/ and /ɑ/ will be subjected to acoustic analysis using TF32 software analyzed for outcome measures 3 and 4.

Focus on vowel assessment was in part because vowels contribute to speech intelligibility. Yet, most formalized speech assessments, including HAPP-3 that we employed, focus predominantly on consonants. Outcome measure 3 was employed for perceptual assessment of vowels. Additionally, vowel acoustic analysis, specifically the first and second formant frequencies (F1 and F2), i.e. the resonant frequencies of the vocal tract, will be used to infer information and gain insight on displacement of articulators, such as tongue advancement-retraction and/or tongue height based on mouth/jaw opening when producing the vowels /æ/ and /ɑ/ (i.e. dimensionality of tongue movement/position). F1 corresponds to tongue height and jaw opening (lower F1 indicates higher tongue position and less jaw opening), while F2 relates to tongue advancement (higher F2 corresponds to a more fronted tongue position). The F2-F1 difference correlates with tongue advancement. Given the complex nature of the speech disorder in DS and the presence of craniofacial anomalies, acoustic modification post intervention - which may not be perceptually salient - could provide insight on the effectiveness of vowel-focused intervention on speech intelligibility despite craniofacial anomalies.

III. The Script program is a motor training treatment guidance. Script templates are common conversational topics with short phrase level productions that are practiced in unison, with prompting (fading unison), and then independently. The script training with visual support aims to improve the motor production/planning of vowels /ɑ/ and /æ/ in sentences while supporting the learning style of individuals with cognitive disabilities. Additionally, productions with variable communication partners may aid generalization. Script topics choices will include a conversation starter, ordering at a restaurant, movie or video game (favorite parts) description, and/or how to invite a friend over. One script will be used per treatment session to practice the production of /ɑ/ and /æ/ vowel contrasts in phrases. Once the vowels are mastered in the initial script, an additional one or two scripts will be chosen by participants and used as home practice. Blocked practice of script phrases motivates their use outside of treatment sessions. To ensure effective intervention, age appropriate activities and materials will be used during treatment while accounting for individual needs and interests. Production of script phrases will be used for outcome measure 6.

IV. Intelligibility in Context Scale is a reliable and valid parent-report tool used for outcome measure 7. It consists of seven items, for parents to rate on a 5-point scale, on how well their child's speech is understood in various social contexts.

The outcome measures listed in the Results will be used to: a) Assess the efficacy of intervention in improving accuracy of speech production and speech intelligibility; and b) Gain insight on motoric limitations versus anatomic constraints on speech accuracy. Findings from this clinical intervention study are expected to pave the path towards identifying optimal management of speech clarity in speakers with DS and provide the preliminary data needed to bridge the gap towards a clinical trial on functional anatomy as an early intervention strategy to promote speech clarity in young children with DS.

ELIGIBILITY:
Inclusion Criteria:

* Males with a diagnosis of Down syndrome between the ages of 7 and 16 years
* Primary language is English
* Interested in improving their speech intelligibility.
* All participants must consent/assent to participate. As this is a multiple single subject design, services are available to all motivated participants who are willing to commit to the time/durations described in the diagnostic treatment.

Exclusion Criteria:

* Primary language is not American English
* Do not have a diagnosis of Down syndrome
* Female
* Ages birth-6 and 17 years or older
* Individuals who have a co-occurring diagnosis that affects communication abilities [e.g., diagnosed as deaf with cochlear implants, Autism, only use an alternative/augmentative communication (AAC) device to communicate],
* Severe hearing loss which will limit their ability to participate in the treatment

  * Individuals with a known mild or moderate hearing loss or current speech- language therapy services will not be excluded, but this information will be requested in the Parent Questionnaire. In addition, access to their current individualized education program (IEP) will be requested.

Ages: 7 Years to 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — At this time, only males are eligible to participate.
Enrollment: 3 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Houri K Vorperian, PhD, CCC-SLP, Principal Investigator — University of Wisconsin, Madison - Waisman Center
Locations (1):
- Waisman Center, 1500 Highland Avenue, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wild A, Vorperian HK, Kent RD, Bolt DM, Austin D. Single-Word Speech Intelligibility in Children and Adults With Down Syndrome. Am J Speech Lang Pathol. 2018 Feb 6;27(1):222-236. doi: 10.1044/2017_AJSLP-17-0002. PMID 29214307
- [Background] Vorperian HK, Kent RD, Lee Y, Bolt DM. Corner vowels in males and females ages 4 to 20 years: Fundamental and F1-F4 formant frequencies. J Acoust Soc Am. 2019 Nov;146(5):3255. doi: 10.1121/1.5131271. PMID 31795713
- [Background] Kent RD, Eichhorn J, Wilson EM, Suk Y, Bolt DM, Vorperian HK. Auditory-Perceptual Features of Speech in Children and Adults With Down Syndrome: A Speech Profile Analysis. J Speech Lang Hear Res. 2021 Apr 14;64(4):1157-1175. doi: 10.1044/2021_JSLHR-20-00617. Epub 2021 Mar 31. PMID 33789057
- [Background] Vorperian HK, Kent RD, Lee Y, Buhr KA. Vowel Production in Children and Adults With Down Syndrome: Fundamental and Formant Frequencies of the Corner Vowels. J Speech Lang Hear Res. 2023 Apr 12;66(4):1208-1239. doi: 10.1044/2022_JSLHR-22-00510. Epub 2023 Apr 4. PMID 37015000
- [Result] Eichhorn JA, Pearl-Soloman N, Vorperian HK. Treatment for Speech Intelligibility in Children with Down Syndrome: A Pilot Clinical Trial. Poster presented at the 2022 Annual Convention of the American Speech-Language Hearing Association in New Orleans, LA.
- See also: University of Wisconsin, Madison, Waisman Center, Vocal Tract Development Lab — https://web.waisman.wisc.edu/www/vocal/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from September 2019 through approximately March 2020.
Groups:
- Speech Therapy: Direct speech therapy will be provided for a 12 week period with up to three one-hour sessions per week (36 sessions per participant) as tolerated and 30 minutes weekly home practice.
Period: Overall Study
Arm/Group | Speech Therapy
Started | 3
Completed Treatment | 3
1 Month Post-intervention | 2
6 Months Post-intervention | 0
Completed | 0
Not Completed | 3
Not completed — COVID-19 pandemic | 3

BASELINE CHARACTERISTICS:
Groups:
- Speech Therapy: Direct speech therapy will be provided for a 12 week period with up to three one-hour sessions per week.
Arm/Group | Speech Therapy
Number analyzed (Participants) | 3
Age, Continuous [Mean (Full Range); unit: years] | 12.42 [10.17 to 13.83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2
  White-Asian | 1
Region of Enrollment [Number; unit: participants]
  United States | 3
Mean Length of Utterance (MLU) [Mean (Full Range); unit: morphemes per utterance] — MLU is calculated by dividing the number of morphemes by the number of utterances (ideally 100), higher MLU indicates a higher level of language proficiency.
  morphemes per utterance | 2.05 [1.93 to 2.13]
Peabody Picture Vocabulary Test (PPVT) [Mean (Full Range); unit: score on a scale] — PPVT is scored between 20-160. 20-69 is an extremely low receptive vocabulary score 70-84 is a moderately low receptive vocabulary score 85-114 is an average receptive vocabulary score
  score on a scale | 78.33 [66 to 88]
Hearing Screening (Pass / Fail) [Count of Participants; unit: Participants] — The American Speech Language Hearing Association criterion for passing a hearing screening is a pure tone average (PTA) from 1000, 2000, and 4000Hz that is better than 30dB Hearing Level in both ears.
  Participants
    Pass | 3
    Fail | 0
Oral Exam: Mouth Posture at Rest [Count of Participants; unit: Participants]
  Open | 2
  Approximated | 1
Oral Exam: Tongue Posture at Rest, In Mouth [Count of Participants; unit: Participants] | 3
Oral Exam: Palate [Count of Participants; unit: Participants]
  High and Narrow | 2
  Refused Exam | 1
Oral Exam: Dental Malocclusion [Count of Participants; unit: Participants] — Class I: The alignment of the teeth is good in general, but there is an abnormal shape to the arch.
  Class II: The upper front teeth alignment is fine, but the lower front teeth lean toward the tongue.
  Class III: The upper arch is underdeveloped.
  Participants
    Class I | 2
    Class II | 0
    Class III | 1
Oral Exam: Orthodontic Treatment [Count of Participants; unit: Participants]
  Palate Expander | 2
  Braces | 1
  None | 1

OUTCOME MEASURES:

1. Primary Outcome: Hodson Assessment of Phonological Patterns-3 (HAPP-3) Occurrence Scores
Description: The HAPP-3 test is designed to assess the phonological disorder severity in children, guide intervention and document progress. This 50-word test categorizes phonological deviations into two patterns to guide intervention: 1) Word/Syllable Structure Omissions (129 total instances): including omission of syllables, consonant clusters, and single consonants; 2) Consonant Category Deficiencies (144 instances): including consonant substitutions and assimilations. The range of the combined sum of errors from both patterns, or the Total Occurrence of Major Phonological Deviations (TOMPD) score, is 0-273 with a severity of phonological disorder rating of 0-150 (0: No errors; 1-50: Mild; 51-100: Moderate; 101-150: Severe; >150: Profound). Lower TOMPD scores imply fewer errors and better speech intelligibility, and higher scores indicate more errors and reduced intelligibility. A decrease in TOMPD score post intervention implicates improvement in speech production.
Time Frame: Baseline (pre-treatment), post-treatment (12 weeks), 1-month post-treatment (16weeks), and 6 months post-treatment (36 weeks)
Population: Individual participant data reported. Only 2 participants (Participant 1 and Participant 3) had a 1 month post-treatment follow up, and data was collected from 0 participants at 6 month post-treatment due to COVID-19 pandemic.
Measure: Number; unit: sum of errors
Groups:
- Speech Therapy - Participant 1; Speech Therapy - Participant 2; Speech Therapy - Participant 3: Direct speech therapy will be provided for a 12 week period with up to three one-hour sessions per week.
Arm/Group | Speech Therapy - Participant 1 | Speech Therapy - Participant 2 | Speech Therapy - Participant 3
Number analyzed (Participants) | 1 | 1 | 1
sum of errors
  Pre-Treatment TOMPD | 21 | 34 | 22
  Post-Treatment TOMPD | 6 | 17 | 11
  Post-Treatment 1 Month Follow Up TOMPD: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up TOMPD | 8 |  | 17
  Pre-Treatment Word/Syllable Omissions Sum | 5 | 5 | 4
  Post-Treatment Word/Syllable Omissions Sum | 2 | 2 | 3
  Post-Treatment 1 Month Follow Up Word/Syllable Omissions Sum: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up Word/Syllable Omissions Sum | 1 |  | 3
  Pre-Treatment Consonant Category Deficiencies Sum | 16 | 29 | 18
  Post-Treatment Consonant Category Deficiencies Sum | 4 | 17 | 8
  Post-Treatment 1 Month Follow Up Consonant Category Deficiencies Sum: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up Consonant Category Deficiencies Sum | 7 |  | 14

2. Primary Outcome: Percentages of the Top 3 Major Phonological Deviations of HAPP-3 Addressed in Intervention
Description: The HAPP-3 Comprehensive Phonological Evaluation Record Form specifies, for each phonological deviation pattern, the number of instances the 50-words contain the various deviation types. For example, 1) Word/Syllable Structure Omissions include 39 Consonant Clusters and 16 Syllables; 2) Consonant Category Deficiencies include 19 Liquids /r, l/ and 42 Stridents /s, f/. This enables the calculation of 'Percent of Occurrence' for each error type, allowing personalized intervention where each speaker's deficiencies with higher percentages are targeted first, using the Cycles phonological approach. Here, the top three occurrences of major phonological deviations and deficiencies that were addressed during intervention are reported: Deficiencies of Liquids and Stridents (for all participants), omission of Consonant Clusters for participants 1 and 3, and omission of Syllables for participant 2. Decrease in percent occurrence post-treatment signifies improvement in phonological skills.
Time Frame: Baseline (pre-treatment), post-treatment (12 weeks), 1 month post-treatment (16 weeks), and 6 months post-treatment (36 weeks)
Population: Individual participant data reported. Only 2 participants had a 1 month post-treatment follow up, and data was collected from 0 participants at 6 month post-treatment due to COVID-19 pandemic.
Measure: Number; unit: percentage of deficient word productions
Arm/Group | Speech Therapy - Participant 1 | Speech Therapy - Participant 2 | Speech Therapy - Participant 3
Number analyzed (Participants) | 1 | 1 | 1
percentage of deficient word productions
  Pre-Treatment Liquids total percentage | 52.6 | 31.58 | 47.37
  Post-Treatment Liquids total percentage | 5.26 | 15.79 | 15.79
  Post-Treatment 1 Month Follow Up Liquids total percentage: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up Liquids total percentage | 10.53 |  | 31.58
  Pre-Treatment Stridents total percentage | 14.29 | 26.19 | 16.67
  Post-Treatment Stridents total percentage | 4.76 | 16.66 | 11.9
  Post-Treatment 1 Month Follow Up Stridents total percentage: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up Stridents total percentage | 9.52 |  | 7.14
  Pre-Treatment Word/Syllable Structures Omissions percentage | 12.8 | 18.75 | 7.69
  Post-Treatment Word/Syllable Structures Omissions percentage | 5.13 | 0 | 5.13
  Post-Treatment 1 Month Word/Syllable Structures Omissions percentage: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Word/Syllable Structures Omissions percentage | 2.56 |  | 7.69

3. Primary Outcome: Pre- and Post-Intervention Percentage of Words and Vowels Correctly Identified by Naïve Listeners in Perceptual Ratings of Vocal Tract Development Lab (VTLab) Stimuli
Description: Two adult naïve listeners will orthographically transcribe participants' speech recordings of VTLab stimuli to assess word and vowel intelligibility. These stimuli, designed for lifespan studies of vowel acoustics, were chosen due to the lack of standardized speech samples for clinical assessment and the predominant focus of most formal tests on consonants, despite vowels' contribution to intelligibility. VTLab stimuli consist of 25 monosyllabic words, including five words each for four extreme vowels (/i, u, æ, ɑ/) and the central vowel (/ə/) as in 'eat', 'hoot', 'hat', 'hot', and 'hug'. Intelligibility is measured by comparing transcriptions to intended target words and calculating the percentage correct for total words, all aforementioned vowels, and the extreme front-back low vowels (/æ/ and /ɑ/), which are reportedly more difficult to produce in speakers with Down syndrome. An increase in correct percentages indicates improved speech intelligibility.
Time Frame: as for outcome 2
Population: Individual participant data reported. Two participants (Participant 1 and Participant 3) had only one of the three baseline recordings; but they had 1 month post-treatment recordings (twice for Participant 1, and once for Participant 3). No participant had 6-month post-treatment recordings due to the COVID-19 pandemic. The overall number of units is unique to the analysis at each time point, as specified in the row title.
Measure: Mean (Full Range); unit: percentage correct
Units Other Than Participants: words/vowels * recordings * listener
Arm/Group | Speech Therapy - Participant 1 | Speech Therapy - Participant 2 | Speech Therapy - Participant 3
Number analyzed (Participants) | 1 | 1 | 1
Number analyzed (words/vowels * recordings * listener) | 840 | 840 | 672
percentage correct
  Pre-Treatment Percentage of Words Correct: number analyzed (words/vowels * recordings * listener) | 70 | 210 | 70
  Pre-Treatment Percentage of Words Correct | 92 [88 to 96] | 77.5 [76 to 79] | 70 [68 to 72]
  Post-Treatment Percentage of Words Correct: number analyzed (words/vowels * recordings * listener) | 140 | 140 | 140
  Post-Treatment Percentage of Words Correct | 62.5 [58 to 67] | 82.5 [80 to 85] | 56.5 [50 to 63]
  Post-Treatment 1 Month Follow Up Percentage of Words Correct: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up Percentage of Words Correct: number analyzed (words/vowels * recordings * listener) | 140 | 0 | 70
  Post-Treatment 1 Month Follow Up Percentage of Words Correct | 75 [74 to 76] |  | 46 [46 to 46]
  Pre-Treatment Percentage of all Vowels Correct: number analyzed (words/vowels * recordings * listener) | 70 | 210 | 70
  Pre-Treatment Percentage of all Vowels Correct | 98 [96 to 100] | 88 [88 to 88] | 80 [80 to 80]
  Post-Treatment Percentage of all Vowels Correct: number analyzed (words/vowels * recordings * listener) | 140 | 140 | 140
  Post-Treatment Percentage of all Vowels Correct | 84 [83 to 85] | 91 [91 to 91] | 72 [70 to 74]
  Post-Treatment 1 Month Follow Up Percentage of Vowels Correct: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up Percentage of Vowels Correct: number analyzed (words/vowels * recordings * listener) | 140 | 0 | 70
  Post-Treatment 1 Month Follow Up Percentage of Vowels Correct | 88 [88 to 88] |  | 69 [62 to 75]
  Pre-Treatment Percentage Vowel /æ/ Correct: number analyzed (words/vowels * recordings * listener) | 14 | 42 | 14
  Pre-Treatment Percentage Vowel /æ/ Correct | 90 [80 to 100] | 84 [80 to 88] | 60 [40 to 80]
  Post-Treatment Percentage Vowel /æ/ Correct: number analyzed (words/vowels * recordings * listener) | 28 | 28 | 28
  Post-Treatment Percentage Vowel /æ/ Correct | 90 [80 to 100] | 100 [100 to 100] | 55 [50 to 60]
  1 Month follow-up Post-Treatment Percentage Vowel /æ/ Correct: number analyzed (Participants) | 1 | 0 | 1
  1 Month follow-up Post-Treatment Percentage Vowel /æ/ Correct: number analyzed (words/vowels * recordings * listener) | 28 | 0 | 14
  1 Month follow-up Post-Treatment Percentage Vowel /æ/ Correct | 90 [80 to 100] |  | 30 [0 to 60]
  Pre-Treatment Percentage Vowel /ɑ/ Correct: number analyzed (words/vowels * recordings * listener) | 14 | 42 | 14
  Pre-Treatment Percentage Vowel /ɑ/ Correct | 100 [100 to 100] | 75 [70 to 80] | 70 [60 to 80]
  Post-Treatment Percentage Vowel /ɑ/ Correct: number analyzed (words/vowels * recordings * listener) | 28 | 28 | 28
  Post-Treatment Percentage Vowel /ɑ/ Correct | 72.5 [70 to 75] | 75 [70 to 80] | 55 [50 to 60]
  1 Month follow-up Post-Treatment Percentage Vowel /ɑ/ Correct: number analyzed (Participants) | 1 | 0 | 1
  1 Month follow-up Post-Treatment Percentage Vowel /ɑ/ Correct: number analyzed (words/vowels * recordings * listener) | 28 | 0 | 14
  1 Month follow-up Post-Treatment Percentage Vowel /ɑ/ Correct | 60 [50 to 70] |  | 60 [40 to 80]

4. Primary Outcome: Pre- and Post-Intervention Vowel Formant Frequencies F1 and F2 for /ɑ/ and /æ/ in Recorded Productions of VTLab Stimuli
Description: The vowel portion of the VTLab word stimuli was analyzed acoustically. Pre- and post-intervention formant frequencies F1 and F2 of seven words per vowel /æ/ and /ɑ/ are reported here, as the intervention provided practice for their distinct front-back productions. F1 and F2 are critical for determining vowel type and specify acoustic space that is related to speech intelligibility, serving as a proxy for articulatory working space (i.e. reflecting dimensionality of tongue movement/position). See Detailed Description section for additional information. Reported here are formant frequencies averaged across all pre- and post-conditions, a feasible comparison given similarity in the F1 and F2 increase/decrease trend across conditions. The F2-F1 difference correlates with tongue advancement, increasing as the tongue moves forward and decreasing as it retracts.
Time Frame: Baseline (pre-treatment), post-treatment (12 weeks)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Hz
Units Other Than Participants: vowels times recordings
Groups:
- Speech Therapy: Participant 1; Speech Therapy: Participant 2; Speech Therapy: Participant 3: Direct speech therapy will be provided for a 12 week period with up to three one-hour sessions per week.
Arm/Group | Speech Therapy: Participant 1 | Speech Therapy: Participant 2 | Speech Therapy: Participant 3
Number analyzed (Participants) | 1 | 1 | 1
Number analyzed (vowels times recordings) | 140 | 140 | 112
Hz
  /æ/ F1 Pre-treatment: number analyzed (vowels times recordings) | 7 | 21 | 7
  /æ/ F1 Pre-treatment | 1064.50 (145.73) | 713.32 (167.12) | 758.14 (45.13)
  /æ/ F2 Pre-treatment: number analyzed (vowels times recordings) | 7 | 21 | 7
  /æ/ F2 Pre-treatment | 2206.13 (129.42) | 2290.79 (239.10) | 2290.71 (150.88)
  /æ/ F1 Post-treatment: number analyzed (vowels times recordings) | 28 | 14 | 21
  /æ/ F1 Post-treatment | 975.75 (166.89) | 829.75 (148.42) | 707.90 (56.85)
  /æ/ F2 Post-treatment: number analyzed (vowels times recordings) | 28 | 14 | 21
  /æ/ F2 Post-treatment | 2289.46 (150.52) | 2191.67 (220.24) | 2058.10 (120.61)
  /ɑ/ F1 Pre-treatment: number analyzed (vowels times recordings) | 7 | 21 | 7
  /ɑ/ F1 Pre-treatment | 1188.14 (115.94) | 1049.33 (100.79) | 821.14 (56.56)
  /ɑ/ F2 Pre-treatment: number analyzed (vowels times recordings) | 7 | 21 | 7
  /ɑ/ F2 Pre-treatment | 1671.29 (172.57) | 1458.58 (148.02) | 1415.14 (157.77)
  /ɑ/ F1 Post-treatment: number analyzed (vowels times recordings) | 28 | 14 | 21
  /ɑ/ F1 Post-treatment | 1209.64 (121.80) | 1013.2 (81.49) | 872.06 (135.75)
  /ɑ/ F2 Post-treatment: number analyzed (vowels times recordings) | 28 | 14 | 21
  /ɑ/ F2 Post-treatment | 1764.43 (165.77) | 1451.93 (130.13) | 1480.11 (181.02)

5. Secondary Outcome: Percentage of the HAPP-3 50-Word Stimuli With Correct Phonetic Transcriptions by Trained Listeners Using the International Phonetic Alphabet (IPA)
Description: Listeners with linguistic training will use the International Phonetic Alphabet (IPA) to phonetically transcribe participants' productions of the Hodson Assessment of Phonological Patterns-3 (HAPP-3) stimuli. The stimuli consist of the 50 test words for phonological deviations analysis, and 12 multisyllabic screening words. The percentage of correct words is calculated by comparing the listeners' transcriptions of the speakers' productions against the transcriptions of the intended target words, then multiplying the ratio by 100. This process is applied separately for the 50 test words and 12 multisyllabic screening words. Transcriptions were completed by three trained listeners: one highly experienced listener and two listeners in-training. Findings from the experienced listener are reported since the pattern of transcription accuracy were similar across all listeners.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: percentage correct
Arm/Group | Speech Therapy - Participant 1 | Speech Therapy - Participant 2 | Speech Therapy - Participant 3
Number analyzed (Participants) | 1 | 1 | 1
percentage correct
  Pre-Treatment percentage total words correct | 31 | 23 | 24
  Post-Treatment percentage total words correct | 53 | 51 | 56
  Post-Treatment 1 Month Follow Up percentage total words correct: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up percentage total words correct | 63 |  | 48
  Pre-Treatment percentage monosyllabic words correct | 35 | 28 | 28
  Post-Treatment percentage monosyllabic words correct | 60 | 61 | 62
  Post-Treatment 1 Month Follow Up percentage monosyllabic words correct: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up percentage monosyllabic words correct | 70 |  | 52
  Pre-Treatment percentage multisyllabic words correct | 17 | 0 | 8
  Post-Treatment percentage multisyllabic words correct | 25 | 83 | 33
  Post-Treatment 1 Month Follow Up percentage multisyllabic words correct: number analyzed (Participants) | 1 | 0 | 1
  Post-Treatment 1 Month Follow Up percentage multisyllabic words correct | 33 |  | 33

6. Secondary Outcome: Number of Scripts Produced
Description: The participants will learn basic Scripts using common communication topics of their choice, such as ordering in a restaurant, discussing their favorite movie, or inviting a friend over. Scripts is a guided motor-training protocol used in speech therapy to improve verbal communication skills in everyday situations. Script templates consist of common conversational topics with short, functional, and personally relevant phrases. They are practiced using a cueing hierarchy: 1) Phrase repetition; 2) Phrase repetition in unison using auditory and visual cues; 3) Phrase repetition with prompting, which involves fading unison through a gradual sequential decrease in auditory and visual cues, including the clinician mouthing words; and 4) Independent production without visual cues. Each participant will practice a total of 3-9 scripts with approximately 4-5 words each (e.g. Do you want to play?). Assessment compares three script productions to target scripts for word order and word count.
Time Frame: during treatment, up to12 weeks
Population: Individual participant data reported.
Measure: Count of Units; unit: script phrase
Units Other Than Participants: script phrase
Arm/Group | Speech Therapy: Participant 1 | Speech Therapy: Participant 2 | Speech Therapy: Participant 3
Number analyzed (Participants) | 1 | 1 | 1
Number analyzed (script phrase) | 3 | 3 | 3
script phrase
  Practiced in Unison | 3 | 3 | 0
  Practiced With Prompting (fading unison) | 3 | 3 | 3
  Practiced Independently | 2 | 2 | 1
  Produced Independently | 0 | 2 | 0

7. Secondary Outcome: Scores for the Intelligibility in Context Scale as Rated by Parent
Description: The Intelligibility in Context Scale is a quick parent reported measure of children's intelligibility. The 7-item questionnaire rates the degree to which children's speech is understood by different communication partners (parents, immediate family, extended family, friends, acquaintances, teachers, and strangers) on a 5-point scale. The score ranges from 7-35, higher scores correlate with higher intelligibility.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number; unit: score on a scale
Arm/Group | Speech Therapy: Participant 1 | Speech Therapy: Participant 2 | Speech Therapy: Participant 3
Number analyzed (Participants) | 1 | 1 | 1
score on a scale
  Pre-treatment | 28 | 19 | 26
  Post-treatment | 28 | 24 | 25
  Post-treatment (1 month follow up): number analyzed (Participants) | 1 | 0 | 1
  Post-treatment (1 month follow up) | 29 |  | 25
  Post-treatment (6 month follow up): number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: through 12 weeks of intensive therapy and follow up visits (up to 5 months on study)
Arm/Group | Speech Therapy
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Speech Therapy (N=3)
Decrease in Speech Intelligibility (Congenital, familial and genetic disorders) | 1 — One participant was tired after a full day at school and full participation in tasks could not be secured.

LIMITATIONS AND CAVEATS:
COVID-19 pandemic-related study termination limited enrollment and hindered our ability to address initial study challenges of obtaining multiple baseline measures for two participants, 1-month post-intervention assessment for another, and 6-month post for all participants. Also, rescheduling the final assessment for the third participant was not possible given fatigue-related behavioral issues. Individualized single-subject design intervention is optimal given individual differences in DS.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-23): https://cdn.clinicaltrials.gov/large-docs/54/NCT04059354/Prot_SAP_000.pdf